CLINICAL TRIAL: NCT00697814
Title: Recovery of Gonadal Function by Clomiphene in Males With Prolactinomas and Persistent Hypogonadism
Brief Title: Clomiphene in Males With Prolactinomas and Persistent Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Julio Abucham, Neuroendocrine Unit
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 1374/04
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Hypogonadotropic Hypogonadism; Prolactinoma
Keywords: Hypogonadotropic hypogonadism; Prolactinoma
MeSH Terms: conditions — Hypogonadism; Prolactinoma | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clomiphene (Experimental): Clomiphene 50 mg/day for 12 weeks
  Interventions: Drug: Clomiphene citrate

INTERVENTIONS:
Drug: Clomiphene citrate — Clomiphene 50 mg/day for 12 weeks

SUMMARY:
Prolactinomas are usually associated with hypogonadotropic hypogonadism in both sexes. Clomiphene citrate is a well known selective estrogen receptor modulator that increases gonadotropin secretion via hypothalamic-pituitary action. We conducted a prospective, open label clinical trial of CC to evaluate its effects in reverting persistent HH in male patients with prolactinomas under dopaminergic agonist treatment.

ELIGIBILITY:
Inclusion Criteria:

* a minimum follow-up of 6 months under DA therapy with normal serum prolactin or with maximum DA dose (3.5 mg/week of cabergoline or 10 mg/day of bromocriptine for at least 2 months)
* serum total testosterone less than 300ng/dl with normal or low LH and FSH levels after discontinuing testosterone replacement for at least 2 months.

Exclusion Criteria:

* impossibility to attend scheduled visits and irregular compliance to DA treatment.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
assess the effects of CC treatment on testosterone levels in male patients with prolactinomas and persistent HH on dopaminergic agonist therapy | 10 days, 4, 8 and 12 weeks

SECONDARY OUTCOMES:
Assess the effects of CC on sexual function, fertility, body composition, lipid and glucose metabolism, and quality of life were also evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Abucham, MD, PhD, Study Chair — Neuroendocrine Unit
Locations (1):
- Neuroendocrine Unit - Escola Paulista de Medicina (UNIFESP), São Paulo, São Paulo, Brazil